CLINICAL TRIAL: NCT05325528
Title: An Exploratory Study of Tislelizumab in Combination With Oxaliplatin and Tegafur for the Treatment of Gastric Cancer With Liver Metastases
Brief Title: Study of Tislelizumab in Combination With SOX for the Treatment of Gastric Cancer With Liver Metastases
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian Chen, Head of Gastrointestinal Surgery, Second affiliated hospital of Zhejiang university School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRWC_GC_I001
Record Dates: First submitted 2022-03-21; First posted 2022-04-13 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Liver Metastases
Keywords: gastric cancer; immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): patients in this arm will be treated with Tislelizumab in Combination with Oxaliplatin and Tegafur
  Interventions: Drug: Tislelizumab in Combination with Oxaliplatin and Tegafur

INTERVENTIONS:
Drug: Tislelizumab in Combination with Oxaliplatin and Tegafur — 6 cycles of Tislelizumab plus SOX regimen every 21 days

SUMMARY:
Liver metastases are one of the most common sites of metastasis in advanced gastric cancer. Chemotherapy remains the mainstay of treatment for these patients, but combination chemotherapy has encountered a bottleneck in improving patient survival, with no significant improvement in survival rates at 1, 3 or 5 years. In a previous phase II clinical study we not only observed the survival benefits of Tislelizumab in the treatment of GI tumors such as liver, oesophageal and some gastric cancers, but also confirmed the safety of Tislelizumab in the treatment of advanced GI tumors. This study is a clinical study of PD-1 monoclonal antibody (Tislelizumab) in combination with SOX (Tegafur + Oxaliplatin) for the treatment of liver metastases from gastric cancer. It aims to further explore a new combination therapy for liver metastases from gastric cancer, which is safe and effective for patients with difficult-to-treat disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (Siewert type II or III)
* Presence of clearly measurable (meeting RECIST 1.1 criteria) liver metastases on imaging assessment and no more than three metastases with a maximum individual diameter of no more than 5 cm
* No previous systemic treatment for advanced or metastatic gastric cancer
* Age 18 - 75 years old
* Eastern Cooperative Oncology Group physical status score of 0 or 1
* Laboratory Tests Tolerant of Chemotherapy
* Hematological Examination: no obvious signs of haematological disease, ANC ≥ 1.5 × 10^9/L, platelet count ≥ 80 × 10^9/L, Hb ≥ 90 g/L, WBC ≥ 3.0 × 10^9/L prior to enrolment and no bleeding tendency
* Biochemical examination: total bilirubin < 1.5 times the upper limit of normal, AST and ALT < 2.5 times the upper limit of normal, creatinine < 1.5 times the upper limit of normal

Exclusion Criteria:

* Other pathological type of tumor
* Presence of metastases to organs other than the liver
* Pregnant or lactating women
* Those with a history of other malignant neoplastic disease in the last 5 years
* those with a history of uncontrolled epilepsy, central nervous system disease or psychiatric disorder, where the investigator will determine whether the clinical severity prevents the signing of an informed consent or affects the patient's compliance with oral medication;
* Clinically severe (i.e. active) heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or arrhythmias requiring pharmacological intervention, or a history of myocardial infarction within the last 12 months
* Have severe diabetes-related complications, such as diabetic nephropathy, diabetic ketosis, etc
* Those with digestive tract obstruction or physiological abnormalities, or suffering from malabsorption syndrome, which may affect the absorption of S-1
* Those who have had gastrointestinal bleeding in the last two weeks, or are at high risk of bleeding as judged by the investigator
* Known to have peripheral nerve disease ≥ NCI-CTC AE grade 1. but with deep tendon reflexes (DTR) only
* Those requiring immunosuppressive therapy for organ transplantation
* Presence of any active, known or suspected autoimmune disease
* Those with uncontrolled severe infections, or other severe concomitant diseases
* Those with hypersensitivity to S-1, Oxaliplatin, Tislelizumab or any of the study drug components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | about 6 months after the enrollment
  The percentage of people in the study who have a partial or complete response to the treatment after 6 cycles of Tislelizumab +Tegafur + Oxaliplatin, according to RECIST1.1

SECONDARY OUTCOMES:
progression-free survival | up to 12 months after the end of last cycle of treatment
  The length of time during and after the treatment, that liver metastasis does not get bigger or present new sites of metastasis, according to RECIST1.1

CONTACTS AND LOCATIONS:
Locations (1):
- gastrointestinal department of second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No